CLINICAL TRIAL: NCT03300141
Title: Bimanual Balanced Reaching With Visual Biofeedback
Brief Title: Looking Glass: Bimanual Balanced Reaching With Visual Biofeedback
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Co-Director, Robotics Laboratory, Arms and Hands Lab, Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00204661
Record Dates: First submitted 2017-09-13; First posted 2017-10-03 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Stroke, Acute; Healthy
Keywords: Upper Extremity; Rehabilitation; Arm; Robotics; Stroke Rehabilitation; Virtual Reality Thearpy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy (Active Comparator): Healthy participants will participate in reaching activity using the Looking Glass and Leap motion tracking system
  Interventions: Other: Healthy Comparative Reaching Task
- Chronic Veridical Visual Feedback (Experimental): Reaching while sitting at the Looking Glass system. The representation of arm movements will directly reflect the participants actual arm movements.
  Interventions: Other: Veridical Visual Feedback
- Chronic Augmented Visual Feedback (Experimental): Reaching while sitting at the Looking Glass system. The representation of a participant's arm movements will be augmented to encourage different movement patterns and improved movement.
  Interventions: Other: Augmented Visual Feedback
- Acute Veridical Visual Feedback (Experimental): Reaching while sitting at the Looking Glass system. The representation of arm movements will directly reflect the participants actual arm movements.
  Interventions: Other: Veridical Visual Feedback
- Acute Augmented Visual Feedback (Experimental): Reaching while sitting at the Looking Glass system. The representation of a participant's arm movements will be augmented to encourage different movement patterns and improved movement.
  Interventions: Other: Augmented Visual Feedback

INTERVENTIONS:
Other: Veridical Visual Feedback — Reaching while sitting at the Looking Glass system. The representation of arm movements will directly reflect the participants actual arm movements.
  Other Names: Reaching
  Arms: Acute Veridical Visual Feedback; Chronic Veridical Visual Feedback
Other: Augmented Visual Feedback — Reaching while sitting at the Looking Glass system. The representation of a participant's arm movements will be augmented to encourage different movement patterns and improved movement.
  Other Names: Reaching; Error Augmentation
  Arms: Acute Augmented Visual Feedback; Chronic Augmented Visual Feedback
Other: Healthy Comparative Reaching Task — Reaching while sitting at the Looking Glass system. This will occur over the course of 1 hour.
  Other Names: Healthy Reaching
  Arms: Healthy

SUMMARY:
The goal of this research study is to increase understanding of error augmentation by applying it to visual feedback during motion tracking with a Leap Motion device - a recently developed optical hand tracking tool - and the LookingGlass - a new, portable virtual reality environment.

In conjunction with the Leap, large, three dimensional work spaces can provide an immersive and virtual augmented environment for rehabilitation. Previously, experiments have utilized the Virtual Reality Robotic and Optical Operations Machine (VRROOM) to create such visually immersive environments. The Robotics lab as part of the Arms and Hands Lab on the 22nd floor of the Shirley Ryan Abilitylab has developed a portable version of this system, which is more compact and clinic-compatible. Combining this visual 3D system with the Leap creates a novel, more capable apparatus for studying error augmentation.

This research study will have 3 different arms: 1.) a healthy group of individuals (Healthy Arm), 2.) a group of stroke survivors within 8 months of stroke (Acute Arm), and 3.) a group of stroke survivors that had their stroke more than 8 months ago (Chronic Arm).

Each Arm will use the Leap motion tracker and the Looking Glass to participate in a reaching intervention. The healthy arm will only participate in 1 visit with an intervention with and without error augmented visual feedback. The Acute Arm and the Chronic Arm will both have 2 groups: 1.) Error Augmented Visual Feedback group and 2.) Non-Augmented or Veridical Visual Feedback group.

The Chronic Arm will have a structured intervention and evaluation protocol: Study staff will administer outcome assessments at 3 time points: a.) prior to intervention, b.) post intervention, and c.) 2 months after the conclusion of intervention. Intervention will occur over the span of 6-8 weeks with the goal of 3 1-hour sessions per week.

The Acute Arm will have a less structured intervention that will occur while the participant is an inpatient at Shirley Ryan AbilityLab. Study staff will administer outcome assessments at at least 2 time points: a.) prior to intervention, b.) post intervention just prior to discharge from Shirley Ryan AbilityLab. Between initial and post intervention evaluations, midpoint evaluations will take place at a maximum of once per week if the participant's schedule, activity tolerance, and length of stay allows. Intervention will consist of 1-hour sessions occurring according to the availability of the participant at the rate of no more than 2 sessions in a 24 hour period.

Investigators hope to investigate these questions:

1. Can the movement of healthy individuals be characterized with error augmented visual feedback and veridical visual feedback?
2. Will error augmented visual feedback or veridical visual feedback result in greater movement ability improvement?

   Investigators hypothesize that in the Chronic Arm, those what trained with error-augmented visual feedback will have improved movement ability compared to those who trained with veridical visual feedback.
3. Is treatment with the looking glass and leap system feasible with an inpatient population?

Investigators hypothesize that this treatment will be feasible for an inpatient population.

ELIGIBILITY:
Inclusion Criteria:

* 8 months post stroke
* FMUE 15-50
* Active shoulder and elbow flexion-extension when supported against gravity to accomplish a forward mediolateral and inferior-superior reaching movements of 30 cm

Exclusion Criteria:

* Bilateral paresis
* Severe sensory deficits in the affected limb
* Severe spasticity preventing movement (MAS 4 or greater at elbow)
* Aphasia, cognitive impairment or affective dysfunction that influence ability to participate in the experiment
* Inability to provide informed consent
* Severe current medical problems
* Diffuse/multiple lesion sites or multiple strokes
* Hemi-spatial neglect or visual field cut preventing subjects from seeing the target
* Inability to maintain the testing positions
* Botox injections in the affected Upper Extremity within the past 4 months
* Concurrent participation in Upper Extremity rehab (research or prescribed therapy)
* Participation in previous, similar robotics intervention studies
* Pregnant women, children and teenagers, prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Score: Pre to Post/Discharge - Chronic and Acute Arms | 1-3 weeks for acute arm; 9 weeks for chronic arm
  Change in Fugl Meyer score from pre-evaluation to post -evaluation

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Score: Pre to Follow-up | 4.5 months
  Change in Fugl Meyer score from pre-evaluation to follow-up-evaluation - Chronic Arm
Amount of use | 1-3 weeks, on average
  Time spent in treatment - Acute Arm
Action Research Arm Test Score: Pre to Post | 1-3 weeks for acute arm; 9 weeks for chronic arm
  Change in Action Research Arm Test score from pre-evaluation to post -evaluation: Chronic and Acute Arms
Action Research Arm Test Score: Pre to Follow-Up | 4.5 months
  Change in Action Research Arm Test score from pre-evaluation to Follow-up -evaluation: Chronic Arm

CONTACTS AND LOCATIONS:
Overall Officials: James Patton, Principal Investigator — Shirley Ryan AbilityLab and University of Illinois at Chicago (UIC)
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Celian C, Puzzi T, Verardi M, Olavarria E, Porta F, Pedrocchi A, Patton JL. Does visual error augmentation offer advantages during bimanual therapy in individuals poststroke? A randomized controlled trial. J Int Med Res. 2025 Aug;53(8):3000605251361115. doi: 10.1177/03000605251361115. Epub 2025 Aug 9. PMID 40781976